CLINICAL TRIAL: NCT02058524
Title: A Pilot and Feasibility Study of Fecal Microbiota Transplantation for Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit and enroll eligible subjects.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB13-0212
Record Dates: First submitted 2013-08-27; First posted 2014-02-10 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Fecal Microbiota Transplantation
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fecal microbiota transplantation (Experimental)
  Interventions: Biological: fecal microbiota transplantation

INTERVENTIONS:
Biological: fecal microbiota transplantation
  Other Names: FMT

SUMMARY:
The investigators are conducting an open-label study of fecal microbiota transplantation (FMT) for adult patients with mildly-moderately active ulcerative colitis. In this pilot study the investigators will evaluate the feasibility, safety, and tolerability of a single application of FMT delivered colonoscopically. The investigators will also characterize the impact of FMT on the microbiota of the recipient and determine if it correlates with the microbiota from the FMT donor.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, aged 18-65 years old
* Prior endoscopic confirmation of UC:

Mildly to moderately active UC with Simple Clinical Colitis Activity Index (SCCAI) activity index >4-9

* Failing standard therapy with:

stable doses of 5-ASA >2 weeks; thiopurines >3 months; or is steroid dependent at a dose <20mg/d; (inability to taper off steroid for longer than 1 week)

* Stable medications dose for at least 2 weeks prior to screening and upon entry into trial
* Ability to understand and willingness to sign informed consent document

Exclusion Criteria:

* Diagnosis of Crohn's disease, indeterminate colitis, or proctitis alone
* Severe or fulminate colitis
* Women who are pregnant or nursing
* Patients who are unable to give informed consent
* Patients who are unable or unwilling to undergo colonoscopy
* Patients who have previously undergone FMT
* Patients who have a confirmed malignancy or cancer
* Patients who are immunocompromised
* Treatment within last 12 weeks with cyclosporine, tacrolimus, infliximab, adalimumab, certolizumab, natalizumab, thalidomide
* Antibiotic use within 2-months of start date
* Participation in a clinical trial in the preceding 30 days or simultaneously during this trial
* Probiotic use within 30 days of start date
* Rectal therapy within 14 days of start date
* Decompensated cirrhosis
* Congenital or acquired immunodeficiencies
* Other comorbidities including:

Diabetes mellitus, cancer, systemic lupus, must be able to tolerate conscious sedation with colonoscopy

* Chronic kidney disease as defined by a GFR <60mL/min/1.73m2 (40)
* History of rheumatic heart disease, endocarditis, or valvular disease due to risk of bacteremia.
* Steroid >20mg/day
* Positive screening and confirmatory tests for HIV 1 & 2, Hepatitis A, B, & C, and Syphilis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Comparison of microbiome pre and post transplant | 12 weeks
  We will analyze and compare the microbiome (bacterial populations) present pre- and post- transplant of the recipient. We will also analyze the microbiome of the donor and compare it to the donor microbiome pre- and post-FMT.

SECONDARY OUTCOMES:
Adverse event frequency | 6 months
  Number of patients with reporting adverse events with type and severity of adverse events reported
Tolerance of procedure | day 0 and day 7
  Tolerability of colonoscopic FMT on Day 0 and Day 7 assessed by Tolerability Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Kahn, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States